CLINICAL TRIAL: NCT01117064
Title: Neuromodulation Therapy Device for the Treatment of Sleep Apnea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Dymedix Corporation (Industry)
Responsible Party: Principal Investigator, John G. Park, MD, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 09-006804
Record Dates: First submitted 2010-02-08; First posted 2010-05-05 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep Apnea; OSA; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NMTD adjustment testing (Active Comparator): We will determine effective NMTD device settings for reducing AHI.
  Interventions: Device: Neuromodulation Therapy Device (NMTD)
- CPAP vs NMTD device (Active Comparator): We will randomly assign previously titrated CPAP vs. NMTD to each subject then compare the resultant AHI between the two devices.
  Interventions: Device: Neuromodulation Therapy Device (NMTD)
- NMTD efficacy and tolerability (Active Comparator): Subjects will undergo two sequential nights of PSG with NMTD to evaluate if there is any stimulus-response extinction over time.
  Interventions: Device: Neuromodulation Therapy Device (NMTD)

INTERVENTIONS:
Device: Neuromodulation Therapy Device (NMTD) — Subjects will have an overnight PSG using CPAP (as previously titrated) for half of the night and NMTD the other half (this order will be randomized). we will monitor NMTD's influence on Apnea Hypopnea Index (AHI), sleep architecture, arousal index, and sleep efficiency compared to the same variables during CPAP use
  Arms: CPAP vs NMTD device
Device: Neuromodulation Therapy Device (NMTD) — Subjects will have an overnight PSG using the NMTD. This device detects reduced airflow via a polymer sensor. When such event is detected, a short burst of sound is administered via earphones. We will determine NMTD's operating characteristics for treatment of OSA. The optimal duration of a detected apnea/hypopnea event before NMTD responds must first be determined. Additional adjustable features include sensitivity of respiratory event sensor, as well as pulse duration, frequency, and intensity of the delivered auditory tone. Since independent adjustment of each of the 4 parameters is not feasible, our screening analysis will test two variables at a time to identify which variables most effectively reduce AHI.
  Arms: NMTD adjustment testing
Device: Neuromodulation Therapy Device (NMTD) — Subjects will undergo two sequential nights of PSG with NMTD to evaluate if there is any stimulus-response extinction over time.
  Arms: NMTD efficacy and tolerability

SUMMARY:
We are looking to test a novel device in the treatment of Obstructive Sleep Apnea (OSA). Rather than using positive pressure to open the airways, we are testing a device that delivers an auditory tone to affect neuromodulation. We will test its efficacy in treating OSA while minimizing sleep disturbance. As this device is much less cumbersome to wear, we hope this therapy device will also improve compliance with treatment.

DETAILED DESCRIPTION:
Neuromodulation Therapy Device for the Treatment of Sleep Apnea

Obstructive sleep apnea (OSA) is a common public health problem with severe health consequences that substantially raises the risk of cardiovascular and cerebrovascular death. Continuous positive airway pressure (CPAP) is currently the most effective treatment option, yet up to half of patients fail to tolerate CPAP and require other approaches. Novel treatments offering alternatives to CPAP are thus sorely needed by those suffering from OSA. The Neuromodulation Therapy Device (NMTD) is a novel potential therapy for OSA. The main goal of our project is to evaluate the efficacy, tolerability, and safety of NMTD in patients with OSA.

Hypothesis 1 - The NMTD device is capable of reducing AHI.

OSA severity is indexed by apnea-hypopnea index (AHI), the number of apnea/hypopnea events occurring hourly during sleep. Our first aim is to determine NMTD's operating characteristics for treatment of OSA. The optimal duration of a detected apnea/hypopnea event before NMTD responds must first be determined. Additional adjustable features include sensitivity of respiratory event sensor, as well as pulse duration, frequency, and intensity of the delivered auditory tone. Since independent adjustment of each of the 4 parameters is not feasible, our screening analysis will test two variables at a time to identify which variables most effectively reduce AHI. This will allow for more practical titration during a therapeutic sleep study and more generalizable application of the device.

Hypothesis 2 - Modified NMTD is as effective and tolerable as CPAP in OSA treatment.

Once Aim 1 is complete and effective NMTD settings have been identified, we will initiate a Phase II NMTD trial to assess efficacy and tolerability. The primary outcome variable will be AHI reduction by NMTD compared with CPAP during a repeat polysomnogram (PSG). We will randomly assign previously titrated CPAP vs. NMTD to each subject then compare the resultant AHI between the two devices. Tolerability will also be assessed by sleep efficiency, arousal index, and sleep architecture. While auditory stimuli below 90 dB threshold should not adversely affect sleep architecture and quality,1 intermittent stimuli given during different sleep stages have not been previously assessed. Therefore, we will monitor NMTD's influence on sleep architecture, arousal index, and sleep efficiency compared to the same variables during CPAP use, allowing us to examine whether NMTD affects sleep quality. We will also assess patient preference in using CPAP versus NMTD.

Hypothesis 3 - NMTD will maintain efficacy with repeated use.

Given the brain's plasticity, it is unknown whether the brain may adapt to such repeated auditory stimuli. Constant auditory stimuli may lead to adaptation, resulting in the stimuli being "ignored." NMTD's stimuli, however, are less likely to lead to significant adaptation since they are intermittent and somewhat random, dependent on apneic or hypopneic events. Subjects will undergo two sequential nights of PSG with NMTD to evaluate if there is any stimulus-response extinction over time. In the future, when more devices are available, we will plan on long-term evaluations.

We propose to test this novel device in the treatment of OSA. This device, if successful, will substantially expand the treatment options for OSA by offering an effective alternative to CPAP with the potential for improved treatment compliance.

Plan:

This is a prospective study evaluating the efficacy of the NMTD in the treatment of OSA.

The study is divided into three consecutive phases, representing the three aims. If eligible, participants will be assigned to the phase that is currently being studied.

* One PSG, using the NMTD all night (32 participants)
* One PSG, split between the NMTD and standard CPAP therapy, randomized as to which is first (20 participants)
* Two consecutive PSGs using the NMTD all night (20 participants) to assess stimulus-response extinction over time (20 participants) All participants will complete a questionnaire about their experience with the device.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years or older
* Completed a comprehensive Sleep Medicine evaluation and a standard split-night polysomnogram
* Able to give informed consent
* Confirmed diagnosis of OSA
* Positive airway pressure device naive

Exclusion Criteria:

* Unsuccessful CPAP titration
* Inability to detect screening tone in either ear without the use of hearing aid
* Inability to tolerate a 37 dB tone
* Need for nocturnal oxygen or non-invasive positive pressure ventilation due to hypoventilation/hypercapnia
* Predominantly mixed or central apneas or those who develop complex sleep apnea during the PSG
* Neurologic disorders such as seizure disorder or narcolepsy
* Psychiatric disorders currently not under adequate control
* Need for nurse or other's assistance during the night due to problems of nocturnal confusion, delirium, or other conditions that would preclude the subject from wearing the device all night
* Pregnancy (will be tested)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
We will determine effective device settings on the Neuromodulation Therapy Device (NMTD). | First year

SECONDARY OUTCOMES:
We will compare the modified NMTD's efficacy and tolerability to that of CPAP in treating OSA. | Second year

CONTACTS AND LOCATIONS:
Overall Officials: John G. Park, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States